CLINICAL TRIAL: NCT02605395
Title: Comparative Randomized, Single Dose, Two-way Crossover Open-label Study to Determine the Bioequivalence of Rabeprazole From Raperazole 20mg DR Tabs (GSK, Egypt) and PARIET 20 mg DR Tabs (JANSSEN, EGYPT) After a Single Oral Dose Administration of Each to Healthy Adults Under Fed Conditions
Brief Title: Bioequivalence Study of Raperazole 20mg DR Tabs and PARIET® 20 mg DR Tabs Under Fed Conditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201528
Record Dates: First submitted 2015-05-14; First posted 2015-11-16 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2017-10

CONDITIONS: Gastrointestinal Diseases
Keywords: Bioequivalence; Fed condition; PARIET 20 mg; IDIAZOLE 20mg; Rabeprazole
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A-Idiazole then Pariet (Experimental): Subjects will receive a single oral dose of IDIAZOLE 20mg DR tabs under fed condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of PARIET 20 mg DR tabs under fed condition in treatment period 2.
  Interventions: Drug: IDIAZOLE 20mg DR tabs; Drug: PARIET 20 mg DR tabs
- Group B-Pariet then Idiazole (Experimental): Subjects will receive a single oral dose of PARIET 20 mg DR tabs under fed condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of Idiazole 20mg DR tabs under fed condition in treatment period 2.
  Interventions: Drug: IDIAZOLE 20mg DR tabs; Drug: PARIET 20 mg DR tabs

INTERVENTIONS:
Drug: IDIAZOLE 20mg DR tabs — IDIAZOLE 20mg DR tabs is a delayed-release, enteric-coated tablets containing 20 mg of rabeprazole sodium.
Drug: PARIET 20 mg DR tabs — PARIET 20 mg DR tabs is a delayed-release, enteric-coated tablets containing 20 mg rabeprazole sodium.

SUMMARY:
This is an open-label, randomized, single dose, two-sequence, two-periods crossover study, separated by 7 days washout interval from the first Study Drug Administration. This study is conducted to determine the bioequivalence of Rabeprazole from IDIAZOLE 20mg Delayed-Release (DR) tablets (tabs) and PARIET 20 mg DR tabs after a single oral dose administration of each to healthy adults fed under conditions.

In Period 1, subjects will be randomized to either Idiazole 20mg DR tabs or PARIET 20 mg DR tabs. Following a washout of at least 7 days, subjects will be crossed over in Period 2 to receive the treatment that they did not receive in Period 1.

PARIET is a registered trademark of EISAI Co. Limited.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, age 18 to 55 years, inclusive.
* Body weight within 10 percent of normal range according to the accepted normal values for body mass index (BMI).
* Medical demographics without evidence of clinically significant deviation from normal medical condition.
* Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
* Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

* Subjects with known allergy to the products tested.
* Subjects whose values of BMI were outside the accepted normal ranges.
* Female subjects who were pregnant, nursing or taking birth control pills.
* Medical demographics with evidence of clinically significant deviation from normal medical condition.
* Results of laboratory tests which are clinically significant.
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
* Subject is on a special diet (for example subject is vegetarian).
* Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
* Subject has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
* Subject intends to be hospitalized within 6 weeks after first study drug administration.
* Subjects who, through completion of this study, would have donated more than 500 milliliter (mL) of blood in 7 days, or 750 mL of blood in 30 days, 1000 mL in 90 days, 1250 mL in 120 days, 1500 ml in 180 days, 2000 mL in 270 days, 2500 mL of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-22 (Actual); Primary Completion 2014-03-30 (Actual); Study Completion 2014-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bioequivalence of rabeprazole from Idiazole 20 milligram (mg) tablets and Pariet 20 mg tablets was investigated after single oral dose administration to healthy participants under fed conditions. This study was conducted from 22 March 2014 to 30 March 2014.
Pre-assignment Details: During this study, 74 participants were screened. One participant was excluded for significant variation in laboratory results at screening and three participants voluntarily withdrew before entering in to period 1. Hence, 70 participants were enrolled and randomized in study, and all 70 participants completed both periods of the study.
Groups:
- Pariet 20 mg Followed by Idiazole 20 mg: Eligible participants received a single oral dose of Pariet 20 mg enteric coated tablet in period 1 followed by Idiazole 20 mg gastro-resistant tablets in period 2. Both the treatments were administered under fed condition. Treatment period 1 and period 2 were separated by a 7 days washout period.
- Idiazole 20 mg Followed by Pariet 20 mg: Eligible participants received a single oral dose of Idiazole 20 mg gastro-resistant tablets in period 1 followed by Pariet 20 mg enteric coated tablet in period 2. Both the treatments were administered under fed condition. Treatment period 1 and period 2 were separated by a 7 days washout period.
Period: Period 1, Day 1
Arm/Group | Pariet 20 mg Followed by Idiazole 20 mg | Idiazole 20 mg Followed by Pariet 20 mg
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Washout Period, Day 2 to Day 7
Arm/Group | Pariet 20 mg Followed by Idiazole 20 mg | Idiazole 20 mg Followed by Pariet 20 mg
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Period 2, Day 8
Arm/Group | Pariet 20 mg Followed by Idiazole 20 mg | Idiazole 20 mg Followed by Pariet 20 mg
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Eligible participants received a single oral dose of Pariet 20 mg enteric coated tablets or Idiazole 20 mg gastro-resistant tablets under fed condition in any of the 2 treatment periods. There was a 7 days washout interval between two study drug administration.
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.76 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 70

OUTCOME MEASURES:

1. Primary Outcome: Maximal Measured Plasma Concentration (Cmax) of Rabeprazole
Description: Blood samples were collected for pharmacokinetic analyses in each period at specified time points. Pharmacokinetic parameters of rabeprazole were estimated using standard non-compartmental methods. The Cmax was computed directly from measured data.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 12, 14 and 24 hours post-dose in period 1 and 2
Population: All subject population comprised of all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- Idiazole 20 mg: Eligible participants received a single oral dose of Idiazole 20 mg enteric coated tablets under fed condition in treatment period 1 or 2.
- Pariet 20 mg: Eligible participants received a single dose of Pariet 20 mg gastro-resistant tablets under fed condition in treatment period 1 or 2.
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Nanograms per milliliter | 393.50 (158.60) | 415.83 (179.24)
Statistical Analysis 1: Comparison: Idiazole 20 mg vs Pariet 20 mg; Test type: Equivalence — The confidence intervals of logarithmically transformed ratio (Idiazole/Pariet) for Cmax to be within 80-125% to prove equivalency; Ratio of means = 95.71, 90% CI 2-sided [90.12 to 101.65]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC [0-t]) of Rabeprazole
Description: Blood samples were collected for pharmacokinetic analyses in each period at specified time points. Pharmacokinetic parameters of rabeprazole were estimated using standard non-compartmental methods. AUC (0-t) was calculated from measured data points from time of administration to time of last quantifiable concentration (Clast) by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: All subject population.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Hour*nanograms per milliliter | 812.30 (461.30) | 843.68 (425.21)
Statistical Analysis 1: Comparison: Idiazole 20 mg vs Pariet 20 mg; Test type: Equivalence — The confidence intervals of logarithmically transformed ratio (Idiazole/Pariet) for AUC(0-t) to be within 80-125% to prove equivalency; Ratio of means = 96.50, 90% CI 2-sided [90.02 to 103.44]

3. Primary Outcome: Mean Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC [0 to Infinity]) of Rabeprazole
Description: Blood samples were collected for pharmacokinetic analyses in each period at specified time points. Pharmacokinetic parameters of rabeprazole were estimated using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: All subject population.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Hour*nanograms per milliliter | 798.59 (314.16) | 931.81 (442.17)
Statistical Analysis 1: Comparison: Idiazole 20 mg vs Pariet 20 mg; Test type: Equivalence — The confidence intervals of logarithmically transformed ratio (Idiazole/Pariet) for AUC (0 to infinity) to be within 80-125% to prove equivalency; Ratio of means = 95.69, 90% CI 2-sided [87.06 to 105.17]

4. Secondary Outcome: Mean Time to the Maximum Plasma Concentration (Tmax) of Rabeprazole
Description: Blood samples were collected for pharmacokinetic analysis in each period at specified time points. Pharmacokinetic parameters of Rabeprazole were estimated using standard non-compartmental methods. Tmax was computed directly from the measured data.
Time Frame: as for outcome 1
Population: All subject population.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Hour | 3.93 (1.06) | 3.86 (1.00)

5. Secondary Outcome: Mean Apparent First-order Elimination or Terminal Rate Constant (Ke) of Rabeprazole
Description: Blood samples were collected for pharmacokinetic analysis in each period at specified time points. Pharmacokinetic parameters of Rabeprazole were estimated using standard non-compartmental methods. Ke was derived from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: All subject population
Measure: Mean (Standard Deviation); unit: Per hour
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Per hour | 0.21 (0.14) | 0.16 (0.09)

6. Secondary Outcome: Mean Terminal Half Life (t1/2) of Rabeprazole
Description: Half life is the period of time required for the concentration or amount of drug in the body to be reduced by one-half. Blood samples were collected for pharmacokinetic analysis in each period at specified time points. Pharmacokinetic parameters of Rabeprazole were estimated using standard non-compartmental methods. t1/2 was calculated as: t1/2 = Ln(2) / (-b), where b was obtained as the slope of the linear regression of the Ln-transformed plasma concentrations versus time in the terminal period of the plasma curve.
Time Frame: as for outcome 1
Population: All subject population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Idiazole 20 mg | Pariet 20 mg
Number analyzed (Participants) | 70 | 70
Hour | 4.49 (2.40) | 5.81 (3.08)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to end of the follow-up (24 hours post last blood sample collected for Period 2; Up to 10 days)
Description: All subject population was used for analysis.
Arm/Group | Idiazole 20 mg | Pariet 20 mg
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.